CLINICAL TRIAL: NCT02737137
Title: Monitoring Combining Neurostimulation and Ultrasound Guidance During the Realization of a Peripheral Nerve Block: Value of Objective Measurement of the Pressure of Injection of the Local Anesthetic
Brief Title: Dynamic Multimodal Monitoring for Ultrasound Guided Peripheral Nerve Blockade
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9654; 2015-A01850-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2016-03-01; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-01

CONDITIONS: Orthopedic Surgery
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual measurement by the anesthetist (Other): Monitoring by ultrasound, Neurostimulation and Measurement Manual of the injection pressure of the local anesthetic : Group 1
  Interventions: Procedure: Manual measurement
- Measurement by a pressure gauge (Experimental): Monitoring by ultrasound, Neurostimulation and measurement with a gauge of the injection pressure of the local anesthetic : Group 2
  Interventions: Procedure: Measurement with a gauge

INTERVENTIONS:
Procedure: Manual measurement — Monitoring by ultrasound, Neurostimulation and Measurement Manual of the injection pressure of the local anesthetic
  Other Names: Manual measurement by the anesthetist
  Arms: Manual measurement by the anesthetist
Procedure: Measurement with a gauge — Monitoring by ultrasound, Neurostimulation and measurement with a gauge of the pressure of injection of the local anesthetic
  Other Names: Measured by a pressure gauge
  Arms: Measurement by a pressure gauge

SUMMARY:
In clinical practice, local anesthetic injection pressure monitoring is performed manually or by a pressure transducer according to the availability of the equipment or preferences of clinicians. To date, no comparative study has measured the advantages of this measure during PNB.

The aim of this study is to evaluate injection pressure monitoring in order to reduce the risk of intraneural injection during peripheral nerve blocks

DETAILED DESCRIPTION:
Current recommendations for peripheral nerve block (PNB) procedure advocate combining ultrasound guidance and nerve stimulation.

Despite these different means of identification, nerves contacts and intraneural injection are frequent. Even rare, nerve damage may occur.

The nerve damage may be related to direct trauma with the needle or inadvertent intra-neural injection. High injection pressure of local anesthetic (AL) is an indicator that further characterize the location of the needle in terms of tissue density. In clinical practice, local anesthetic injection pressure monitoring is performed manually or by a pressure transducer according to the availability of the equipment or preferences of clinicians. To date, no comparative study has measured the advantages of this measure during PNB.

The aim of this study is to evaluate injection pressure monitoring in order to reduce the risk of intraneural injection.

Group 1: ultrasound-guided technique PNB "in plane" needle approach, nerve stimulator set to sentinel mode. Manual injection pressure control Group 2: ultrasound-guided PNB, "in plane" approach, Nerve stimulator set to detection mode. Electronic Injection Pressure controlled with low flow local anesthetic during procedure

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Orthopedic surgery

Exclusion Criteria:

* Allergy to local anesthetics
* ASA score >III
* Severe neuropathy
* puncture site disease
* parturient or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Manual measurement | Intraoperative
  Manual measurement of the pressure of injection of the local anesthetic during surgery for patients in Group 1

SECONDARY OUTCOMES:
Measured by a pressure gauge | Intraoperative
  Measured by a pressure gauge of the pressure of injection of the local anesthetic during surgery for patients in Group 2

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHOQUET, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHOQUET, France, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided